CLINICAL TRIAL: NCT01052038
Title: The Effect of Systemic Prophylactic Dexamethasone on the Incidence of Postoperative Sore Throat in Patients Undergoing Ambulatory Laparoscopic Gynecologic Surgery: A Prospective, Randomized, Double Blinded, Placebo Controlled Trial
Brief Title: Post Operative Sore Throat and Dexamethasone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Gildasio De Oliveira, Gildasio De Oliveira, M.D. Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STU00018901
Record Dates: First submitted 2010-01-19; First posted 2010-01-20 (Estimated); Results first posted 2012-05-02 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-04

CONDITIONS: Sore Throat; Pain
Keywords: Sore throat; Dexamethasone; Pain
MeSH Terms: conditions — Pharyngitis; Pain | interventions — Calcium Dobesilate; Adrenal Cortex Hormones; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 Placebo (Placebo Comparator): Normal saline 100ml (placebo) administered as a intravenous infusion 30 minutes prior to surgery.
  Interventions: Drug: Placebo administration
- Group 2: Dexamethasone 0.05mg/kg (Active Comparator): Dexamethasone 0.05 mg/kg administered in 100 ml of sterile saline solution prior to surgery
  Interventions: Drug: Dexamethasone 0.05mg/kr administration
- Group 3:Dexamethasone 0.1mg/kg (Active Comparator): Dexamethasone 0.1mg/kg administered in 100ml of sterile saline solution prior to surgery.
  Interventions: Drug: Dexamethasone 0.1mg/kg

INTERVENTIONS:
Drug: Placebo administration — Placebo administration
  Other Names: Decadron; Corticosteroid
  Arms: Group 1 Placebo
Drug: Dexamethasone 0.05mg/kr administration — Dexamethasone 0.05mg/kr administered in 100ml of sterile saline solution prior to the start of surgery.
  Other Names: Decadron; corticosteroid
  Arms: Group 2: Dexamethasone 0.05mg/kg
Drug: Dexamethasone 0.1mg/kg — Dexamethasone 0.1mg/kg administered in 100ml of sterile saline solution prior to the beginning of surgery.
  Other Names: Decadron; corticosteroid
  Arms: Group 3:Dexamethasone 0.1mg/kg

SUMMARY:
Sore throat is a common postoperative complaint that can lead to morbidity and patient dissatisfaction . The incidence of sore throat has been reported to be between 6% and 90% even under optimal intubating conditions. There are several factors that have been shown to contribute to postoperative sore throat such as patient related factors, type of anesthesia and type of surgery.

Corticosteroids are also commonly used in the perioperative period to potentiate analgesics and as antiemetics. The preoperative administration of dexamethasone can decrease the incidence and severity of postoperative sore throat which is rated by patients as one of the most undesirable outcomes in the postoperative period.

DETAILED DESCRIPTION:
Sore throat is a common postoperative complaint that can lead to morbidity and patient dissatisfaction. The incidence of sore throat has been reported to be between 6% and 90% even under optimal intubating conditions. There are several factors that have been shown to contribute to postoperative sore throat such as patient related factors, type of anesthesia and type of surgery. It has been observed that gargle with azunol reduced the incidence of postoperative sore throat from 65% to 25 %. Similarly, a reduction in sore throat following tracheal intubation from 78% to 40 % has been reported after gargle with ketamine performed 5 minutes before induction of anesthesia. More recently, it was also demonstrated that preoperative gargle with licorice resulted in a 57 percent reduction of the absolute risk of sore throat after intubation. Although the gargling technique has been shown to be successful in decreasing the incidence of postoperative sore throat, it has a limited feasibility because the volumes administered could increase the chance of aspiration if ingested and it may be difficult to perform in sedated patients and in children.

Tracheal intubation is associated with an increase of polymorphonuclear cells in the tracheal tissue and plasma levels of interleukin 6, suggesting an inflammatory response to the presence of the endotracheal tube itself or to some aspect of the intubation process. Dexamethasone is widely prescribed for the treatment of a sore throat resulting from tracheal mechanical irritation due to its modulating effects of tissue edema and pain. Moreover, prophylactic dexamethasone has been shown to be effective in reducing the frequency of airway obstruction in patients at high risk for laryngeal edema following extubation. It decreases postoperative sore throat in patients requiring double-lumen tubes.

Dexamethasone has been shown to decrease postoperative sore throat in patients requiring hospital admission but it has not been evaluated in the ambulatory setting. Ambulatory patients usually need to return to work faster than patients who are admitted to the hospital. Their ability to tolerate fluids and food might help them to return to normal living. They also have smaller surgeries which might increased their perception to sore throat pain when compared to bigger, more painful procedures.

Possible side effects of corticosteroids such as retardation of wound healing, susceptibility to infection and gastrointestinal hemorrhage have not been noted with short term use (<24 hours ) in surgical patients. Corticosteroids are also commonly used in the perioperative period to potentiate analgesics and as antiemetics.

ELIGIBILITY:
Inclusion Criteria:

* Female patients undergoing outpatient laparoscopic gynecologic surgery
* ASA PS I and II
* Age between 18 and 64 years
* Fluent in English

Exclusion Criteria:

* History of recent respiratory tract infection
* Pregnancy, breastfeeding
* Current treatment with analgesics
* Current use of corticosteroids
* Anticipated difficult intubation
* Risk factors for post-operative aspiration

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2010-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gildasio DeOliveira, M.D., Principal Investigator — Northwestern University
Locations (1):
- Northwesten University, Chicago, Illinois, United States

REFERENCES:
- [Result] De Oliveira GS Jr, Ahmad S, Fitzgerald PC, Marcus RJ, Altman CS, Panjwani AS, McCarthy RJ. Dose ranging study on the effect of preoperative dexamethasone on postoperative quality of recovery and opioid consumption after ambulatory gynaecological surgery. Br J Anaesth. 2011 Sep;107(3):362-71. doi: 10.1093/bja/aer156. Epub 2011 Jun 13. PMID 21669954

RESULTS

PARTICIPANT FLOW:
Recruitment Details: ASA physical status I and II females undergoing outpatient gynaecological laparoscopy. Patients with a history of recent respiratory tract infection (<1 month), current use of an opioid analgesic or corticosteroid, pregnancy, or anticipated difficult airways were not enrolled. Subjects were enrolled between January 2010 thru September 2010.
Pre-assignment Details: No subjects were lost or excluded after consent was signed and prior to allocation.
Period: Overall Study
Arm/Group | Group 1 Placebo | Group 2: Dexamethasone 0.05mg/kg | Group 3:Dexamethasone 0.1mg/kg
Started | 40 | 40 | 40
Completed | 36 | 34 | 36
Not Completed | 4 | 6 | 4
Not completed — Lost to Follow-up | 2 | 3 | 1
Not completed — Protocol Violation | 2 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 Placebo | Group 2: Dexamethasone 0.05mg/kg | Group 3:Dexamethasone 0.1mg/kg | Total
Number analyzed (Participants) | 40 | 40 | 40 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 40 | 40 | 40 | 120
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 36 (11) | 36 (7) | 39 (11) | 37 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 40 | 120
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 40 | 120

OUTCOME MEASURES:

1. Primary Outcome: Subjects Assessment of Sore Throat Pain at 24 Hours
Description: The reported score for sore throat on a 1 to 5 scale where 1 is a severe sore throat and 5 is no sore throat. This evaluation was made by investigator initiated phone conversation at 24 hours following surgery.
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: units on a scale (1 to 5)
Arm/Group | Group 1 Placebo | Group 2: Dexamethasone 0.05mg/kg | Group 3:Dexamethasone 0.1mg/kg
Number analyzed (Participants) | 40 | 40 | 40
units on a scale (1 to 5) | 4 [3 to 5] | 4 [3 to 5] | 5 [4 to 5]
Statistical Analysis 1: Comparison: Group 1 Placebo vs Group 2: Dexamethasone 0.05mg/kg vs Group 3:Dexamethasone 0.1mg/kg; Test type: Superiority or Other; p < 0.001, Kruskal-Wallis
Statistical Analysis 2: Comparison: Group 1 Placebo vs Group 3:Dexamethasone 0.1mg/kg; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney); Median Difference (Net) = 1, 95% CI 2-sided [0 to 2]
Statistical Analysis 3: Comparison: Group 2: Dexamethasone 0.05mg/kg vs Group 3:Dexamethasone 0.1mg/kg; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney); Median Difference (Net) = 1, 95% CI 2-sided [0 to 2]

2. Secondary Outcome: Quality of Recovery at 24 Hours
Description: The quality of recovery (QoR-40) questionnaire assess the subjects perceived quality of recovery following surgery. The tool assess pain, physical and psychological well being as well as ability to ability for self-care. Questions are scored on a 1 to 5 point scale with a higher value indication a better outcome. The scores or the individual questions are summed to obtain a total score. The minimum total score is 30 and the maximum is 200. The higher the score the better the recovery
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: units on a scale (30 to 200) higher scod
Arm/Group | Group 1 Placebo | Group 2: Dexamethasone 0.05mg/kg | Group 3:Dexamethasone 0.1mg/kg
Number analyzed (Participants) | 40 | 40 | 40
units on a scale (30 to 200) higher scod | 171 [160 to 182] | 179 [175 to 185] | 193 [192 to 195]
Statistical Analysis 1: Comparison: Group 1 Placebo vs Group 2: Dexamethasone 0.05mg/kg vs Group 3:Dexamethasone 0.1mg/kg; Test type: Superiority or Other; p < 0.001, Kruskal-Wallis; Dunn's post hoc-test corrected for 12 comparisons
Statistical Analysis 2: Comparison: Group 1 Placebo vs Group 3:Dexamethasone 0.1mg/kg; Test type: Superiority or Other; p = 0.005, Wilcoxon (Mann-Whitney); Median Difference (Net) = 22, 95% CI 2-sided [14 to 29]
Statistical Analysis 3: Comparison: Group 2: Dexamethasone 0.05mg/kg vs Group 3:Dexamethasone 0.1mg/kg; Test type: Superiority or Other; p = 0.004, Wilcoxon (Mann-Whitney); Median Difference (Net) = 14, 95% CI 2-sided [7 to 22]

3. Secondary Outcome: Number of Subjects With Sore Throat at 3 Hours Post Surgery.
Description: Subjects were asked at 3 hours post surgery if they were experiencing a sore throat.
Time Frame: 3 hours.
Measure: Number; unit: participants
Arm/Group | Group 1 Placebo | Group 2: Dexamethasone 0.05mg/kg | Group 3:Dexamethasone 0.1mg/kg
Number analyzed (Participants) | 40 | 40 | 40
participants | 24 | 17 | 10
Statistical Analysis 1: Comparison: Group 1 Placebo vs Group 2: Dexamethasone 0.05mg/kg vs Group 3:Dexamethasone 0.1mg/kg; Test type: Superiority or Other; p = 0.004, Chi-squared, Corrected

4. Secondary Outcome: Opioid Consumption at 24 Hours
Description: The cumulative use of an opioid analgesic pain medication taken during the first 24 hours for pain and discomfort. Data reported as equivalent dose of oral morphine.
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: mg of oral morphine equivalents
Arm/Group | Group 1 Placebo | Group 2: Dexamethasone 0.05mg/kg | Group 3:Dexamethasone 0.1mg/kg
Number analyzed (Participants) | 40 | 40 | 40
mg of oral morphine equivalents | 20 [20 to 30] | 20 [10 to 32.5] | 10 [10 to 20]
Statistical Analysis 1: Comparison: Group 1 Placebo vs Group 2: Dexamethasone 0.05mg/kg vs Group 3:Dexamethasone 0.1mg/kg; Test type: Superiority or Other; p = 0.01, Kruskal-Wallis; Post hoc test using Dunn's test corrected for 12 comparisons
Statistical Analysis 2: Comparison: Group 1 Placebo vs Group 3:Dexamethasone 0.1mg/kg; Test type: Superiority or Other; p = 0.003, Wilcoxon (Mann-Whitney); Median Difference (Net) = 10, 95% CI [0 to 20]

5. Secondary Outcome: Hoarseness at 24 Hours
Description: Self assessment of the degree of hoarseness 24 hours after surgery and intratracheal intubation on a 1 to 1 Likert scale. 0 = no hoarseness and 3= hoarseness easily noted at time of interview.
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | Group 1 Placebo | Group 2: Dexamethasone 0.05mg/kg | Group 3:Dexamethasone 0.1mg/kg
Number analyzed (Participants) | 40 | 40 | 40
participants
  No hoarseness | 5 | 11 | 18
  No hoarseness at interview but present during 24h | 10 | 6 | 8
  Hoarseness at interview noted by patient | 15 | 11 | 6
  Hoarseness easily noted by interviewer | 6 | 6 | 4
Statistical Analysis 1: Comparison: Group 1 Placebo vs Group 2: Dexamethasone 0.05mg/kg vs Group 3:Dexamethasone 0.1mg/kg; Test type: Superiority or Other; p = 0.04, Chi-squared, Corrected

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 24 hours following surgery
Arm/Group | Group 1 Placebo | Group 2: Dexamethasone 0.05mg/kg | Group 3:Dexamethasone 0.1mg/kg
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 25/40 | 19/40 | 18/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 Placebo (N=40) | Group 2: Dexamethasone 0.05mg/kg (N=40) | Group 3:Dexamethasone 0.1mg/kg (N=40)
Sore throat (Surgical and medical procedures) | 25 (25) | 19 (19) | 18 (18)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 20 (20) | 3 (3) | 6 (6)
Coughing (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 8 (8) | 6 (6)

LIMITATIONS AND CAVEATS:
Study was limited to 2 doses of dexamethasone and was underpowered to assess side effects such as hyperglycemia or delayed wound healing. Study was limited to a single type of surgery and results may differ in different types of surgery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes